CLINICAL TRIAL: NCT01878019
Title: Mechanisms of Pain Control in Chronic Pain Patients
Brief Title: Brain Response to Pain Control in People With Chronic Pain
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130143; 13-AT-0143
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2016-09-08

CONDITIONS: Pain
Keywords: Pain; Placebo; Opiate Antagonist
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Researchers want to look at how the brain responds to painful stimulations. They also want to see if these responses are different in people with and without chronic pain. To test the brain s response, they will use a chemical called naloxone. Naloxone is used to treat overdoses of painkilling drugs like morphine. It may be able to block the effect of a pain-relieving cream. Researchers will apply a pain-relieving cream to a person s lower leg and look at the results of sensitivity tests with either naloxone or a placebo. This study will compare the results from people with chronic pain (like fibromyalgia) to those of people without chronic pain.

Objectives:

- To look at the brain s response to pain in people with and without chronic pain.

Eligibility:

* Individuals at least 18 years of age who have fibromyalgia.
* Healthy volunteers at least 18 years of age.

Design:

* This study will involve a screening visit and two testing visits. The testing visits will be about a week apart.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. After the screening participants will be administered several questionnaires about their personality, and their thoughts and feelings.
* At the first visit, participants will try out the magnetic resonance imaging (MRI) scan before using it at the next visit. They will then have the painkilling cream applied on one part of their lower leg and a normal moisturizing cream on the other part of their lower leg. They will have heat pulses on these skin areas and rate the pain.
* At the second visit, participants will have tests in the MRI scanner. The heat pulse tests will be repeated after an infusion of either naloxone or a placebo.

DETAILED DESCRIPTION:
Different pain reducing drugs work in different ways to reduce pain. Many drugs, including morphine and codeine, reduce pain by binding to opiate receptors in the brain. Another chemical, naloxone, can block the effect of these drugs. In this study, we are looking at brain responses to a pain-relieving cream and whether naloxone blocks the effect of the cream. We will compare the results of people with chronic pain (fibromyalgia) to those of people without chronic pain.

Design:

The study compares MRI response to painful stimulation between people with fibromyalgia and healthy volunteers under two conditions: 1) naloxone, 2) placebo.

Outcome measures: Pain ratings and pain-related MRI responses are compared between people with fibromyalgia and healthy volunteers

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Patients:

1. Patient must be greater than or equal to 18 years of age.
2. Patient must be able to comprehend English.
3. Patient must be able to provide written informed consent.
4. Patient must have had chronic widespread pain for at least one year prior to participation with an average daily intensity at least 4 out of 10.

Inclusion Criteria for Healthy Controls:

1. Healthy control must be greater than or equal to 18 years of age
2. Healthy control must be able to comprehend English.
3. Healthy control must be able to provide written informed consent.

EXCLUSION CRITERIA:

Exclusion criteria for patients:

1. Patient is unable to comply with study procedures or follow-up visits
2. Patient smokes more than 10 cigarettes of nicotine per week.
3. Patient uses recreational drugs.
4. Female patient consumes more than 7 half-pint beers, 7 6-oz glasses of wine or 7 1-oz shots of spirits (or equivalent) per week, and male patient consumes 14 such drinks per week. Further, patient consumes more than 5 drinks at one time.
5. Patient is pregnant or breastfeeding.
6. Patient has a major medical condition, such as kidney, liver, cardiovascular, neurological or current psychiatric condition.
7. Patient has currently or has had in the past major depression, bipolar disorder, psychosis or suicide attempts.
8. Patient has metal in his/her body which would make having an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have.
9. Patient is uncomfortable in small closed spaces (has claustrophobia) so that he/she would feel uncomfortable in the MRI machine.
10. Patient cannot lie comfortably flat on his/her back for up to 75 minutes in the MRI scanner.
11. Patient has allergies to topical treatment.
12. Patient has a chronic pain condition other than FM.
13. Patient has taken within the last two weeks opioids. Other medications used to treat fibromyalgia at the standard doses in the community can be taken. We will not ask participants to stop any medication to participate in the study.
14. Patient has previously taken opioids for more than one month on a continual basis, within the last 6 months.
15. Patient had seen study information on clinicaltrials.gov prior to September 23, 2013.
16. Patients who decline to be audio and/or videotaped will be excluded from the qualitative interview component of the study.

Exclusion criteria for healthy controls:

1. Healthy control is unable to comply with study procedures or follow-up visits
2. Healthy control smokes more than 10 cigarettes of nicotine per week.
3. Healthy control uses recreational drugs.
4. Female healthy control consumes more than 7 half-pint beers, 7 6-oz glasses of wine or 7 1-oz shots of spirits (or equivalent) per week, and male healthy control consumes 14 such drinks per week. Further, healthy control consumes more than 5 drinks at one time.
5. Healthy control is pregnant or breastfeeding.
6. Healthy control has a major medical condition, such as kidney, liver, cardiovascular, neurological or current psychiatric condition.
7. Healthy control has currently or has had in the past major depression, bipolar disorder, psychosis or suicide attempts.
8. Healthy control has metal in his/her body which would make having an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-05-28; Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Pain Perception | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Bushnell, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Apkarian AV, Sosa Y, Sonty S, Levy RM, Harden RN, Parrish TB, Gitelman DR. Chronic back pain is associated with decreased prefrontal and thalamic gray matter density. J Neurosci. 2004 Nov 17;24(46):10410-5. doi: 10.1523/JNEUROSCI.2541-04.2004. PMID 15548656
- [Background] Atlas LY, Bolger N, Lindquist MA, Wager TD. Brain mediators of predictive cue effects on perceived pain. J Neurosci. 2010 Sep 29;30(39):12964-77. doi: 10.1523/JNEUROSCI.0057-10.2010. PMID 20881115
- [Background] Baliki MN, Geha PY, Fields HL, Apkarian AV. Predicting value of pain and analgesia: nucleus accumbens response to noxious stimuli changes in the presence of chronic pain. Neuron. 2010 Apr 15;66(1):149-60. doi: 10.1016/j.neuron.2010.03.002. PMID 20399736